CLINICAL TRIAL: NCT03344692
Title: Effect of Alirocumab on Postprandial Hyperlipemia in Patients With Type 2 Diabetes : a Randomized, Double-blind, Placebo-controlled, Cross-over Trial"
Brief Title: Effect of Alirocumab on Postprandial Hyperlipemia in Patients With Type 2 Diabetes
Acronym: EUTERPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC16_0406
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alirocumab (Experimental): Alirocumab 75 mg for subcutaneous injection via a pre-filled pen. One injection every 2 weeks during a 10-weeks period (5 injections in total)
  Interventions: Drug: Alirocumab
- Placebo (Placebo Comparator): Placebo matching alirocumab is prepared in the same formulation as alirocumab, without the addition of protein, for subcutaneous injection via a pre-filled pen.
  One injection every 2 weeks during a 10-weeks period (5 injections in total)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alirocumab — prefilled pen containing 75 mg of Praluent (Alirocumab) in 1 ml of solution
  Arms: Alirocumab
Other: Placebo — prefilled pen containing 1 ml of solution without Praluent
  Arms: Placebo

SUMMARY:
Proprotein convertase subtilisin/kexin type 9 (PCSK9) has emerged over the past decade as a post-transcriptional regulator of the LDL receptor (LDL-R). PCSK9 acts as an endogenous natural inhibitor of the LDL-R pathway. Monoclonal antibodies (mAb) directed against PCSK9, such as Alirocumab, are the most common method of PCSK9 inhibition.

The goal of the present study is to assess, in the context of type 2 diabetes, a situation associated with an increased post-prandial hyperlipemia, whether PCSK9 inhibition with Alirocumab affects postprandial intestinal lipoprotein metabolism.

DETAILED DESCRIPTION:
Recently, human monoclonal antibodies directed against PCSK9 have been shown to be effective in reducing LDL cholesterol. Besides the liver, little is known about the role of PCSK9 in the small intestine, a tissue where it is expressed at a high level. Preclinical studies in mice indicate that PCSK9 inhibition reduces post-prandial hyperlipemia.

Here, the investigators will test the effect of PCSK9 inhibition with alirocumab, a PCSK9 mAb, on post-prandial hyperlipemia in 24 patients with type 2 diabetes. The investigators will perform a randomized, double-blind, placebo-controlled, cross-over trial with alirocumab 75 mg every two weeks.

In the cross-over design, two periods of 10-weeks treatment (i.e. 5 injections) will be separated by a 10-week wash-out period to avoid carry-over effect. The primary endpoint will be the total area under the post-prandial triglycerides concentration-time curve from meal-time until 8h (AUC0-8h) after a standardized meal test. As secondary endpoints, the investigators will explore the effect of alirocumab on plasma lipids, markers of cholesterol absorption and synthesis, and glycemic parameters.

This study will help to decipher the function of PCSK9 on intestinal lipoprotein metabolism in human and to determine whether alirocumab can reduce post-prandial hyperlipemia, which is an independent cardiovascular risk factor. From a patient perspective, this study will give some important clues for the management of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Men with type 2 diabetes diagnosed since ≥ 6 months
* HbA1C <9.0%
* Men with primary hypercholesterolemia and/or mixed dyslipidemia
* Aged 18-75 years (limits inclusive)
* Patient could be treated for type 2 diabetes when diet and physical activity are not sufficient to restore glycemic control. The treatment must be stable 1 month before the inclusion and have to remain unchanged all along the study. The only authorized treatments are:
* Metformin
* And/or Sulphonylureas (SUs)
* And/or Repaglinide
* And/or DPP-4 inhibitors
* And/or GLP1 receptor agonists: exenatide, liraglutide, dulaglutide
* Fasting serum TG ≥ 150 mg/dl and < 500 mg/dl
* BMI: 20-45 kg/m2
* Use of statins or ezetimibe is allowed if treatment is stable for ≥ 1 month before the screening

Exclusion Criteria:

* Any secondary causes of hypercholesterolemia or of mixed dyslipidemia (nephrotic syndrome, hypothyroidism…)
* impaired liver function (AST and/or ALT ≥ 3ULN)
* impaired renal function (eGFR with CKD-EPI formula < 30 ml/min)
* Alcohol abuse (> 2 standard alcoholic drink per day; 1 standard alcoholic drink is the equivalent of 10g of alcohol)
* History of myocardial infarction, acute coronary syndrome, unstable angina pectoris, stroke, transient ischemic attack, or cardiac revascularization within the 6 months before the screening visit.
* History of PCSK9 mAb use
* Known sensitivity to monoclonal antibody therapeutics or to their excipients
* Lipid lowering therapies (other than statins), including fibrates, omega-3 fatty acids, bile acid sequestrants, niacin.
* Insulin-treated patients
* History of bariatric surgery
* Inflammatory bowel diseases and gastrointestinal malabsorption diseases
* Uncontrolled hypothyroidism (TSH > ULN and Free T4 < ULN) or hyperthyroidism (TSH < ULN)
* Active cancer: progressive cancer or remission ≤ 3 years, except for basal or squamous cell carcinoma of the skin that has been successfully treated
* Known history of positive test for HIV, hepatitis C or chronic hepatitis B
* Corticosteroids therapy
* Minors
* Adults under guardianship or trusteeship

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Total area under the post-prandial triglycerides concentration-time curve from meal-time until 8h (AUC0-8h) after standardized high fat meal. | During 8 hours at week 10 after first treatment injection
  Fifteenth days after the fifth injection of treatment (thus 10 weeks after first injection of treatment), subjects will be reported to investigational site (after a 12 hours overnight fast). Subjects must consume the test meal within 15 min. Upon completion of the meal (T0), sequential postprandial measurements of triglycerides concentrations will be taken. Blood samples will be collected at T-15, every 30 min for the first two hours after meal consumption, thereafter in 60 min intervals from T120 until 240 min and thereafter in 120 min intervals from T240 until 480 min.

SECONDARY OUTCOMES:
Effect of treatment with alirocumab versus placebo following a standardized high-fat meal on post-prandial lipid metabolism (plasma lipoproteins, apolipoproteins, ...) | During 8 hours at week 10 after first treatment injection
  Fifteenth days after the fifth injection of treatment (thus 10 weeks after first injection of treatment), subjects will be reported to investigational site (after a 12 hours overnight fast). Subjects must consume the test meal within 15 min. Upon completion of the meal (T0), sequential postprandial measurements of triglycerides concentrations will be taken. Bleed samples will be collected at T-15, every 30 min for the first two hours after meal consumption, thereafter in 60 min intervals from T120 until 240 min and thereafter in 120 min intervals from T240 until 480 min.
Effect of treatment with alirocumab versus placebo on fasting lipid metabolism following a standardized high fat meal, using the same biomarkers than those used in the post-prandial state, plus indirect markers of cholesterol absorption and synthesis | 10 weeks after treatment first injection
  Fifteenth days after the fifth injection of treatment (thus 10 weeks after first injection of treatment), subjects will be reported to investigational site after a 12 hours overnight fast. Before ingestion of the high fat meal, blood sample will be removed to perform the analysis.
Effect of treatment with alirocumab versus placebo on fasting and post-prandial and glucose homeostasis following a standardized high-fat meal | Before and during 8 hours after high fat meal at week 10 after first treatment injection
  Fasting self-monitored blood glucose test will be obtained before starting the meal and every hour during 8 hours .

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand CARIOU, Study Chair — Nantes University Hospital
Locations (1):
- University Hospital of Nantes, Nantes, France